CLINICAL TRIAL: NCT01567202
Title: A Triple-blind Randomized Clinical Study of Vaccination With Dendritic Cells Loaded With Glioma Stem-like Cells Associated Antigens Against Brain Glioblastoma Multiform
Brief Title: Study of DC Vaccination Against Glioblastoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: Fudan University (Other)
Responsible Party: Principal Investigator, Jinsong Wu, M.D., Ph.D., Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DC81001115
Record Dates: First submitted 2012-03-26; First posted 2012-03-30 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Glioma; Glioblastoma Multiforme; Neoplasms
Keywords: Brain tumor; Glioma; Glioblastoma; Tumor stem cells; Immunotherapy; Vaccine
MeSH Terms: conditions — Glioma; Glioblastoma; Neoplasms; Brain Neoplasms | interventions — Surgical Procedures, Operative; Drug Therapy; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm DC (Experimental): In this arm, the patients will receive DC vaccination in addition to the standard therapy, including Surgery, Chemotherapy, and Radiotherapy.
  Interventions: Procedure: Surgery; Drug: Chemotherapy; Radiation: Radiotherapy; Biological: DC vaccination
- Arm Placebo (Placebo Comparator): In this arm, the patients will receive blank placebo instead of the DC vaccination in addition to the standard therapy.
  Interventions: Procedure: Surgery; Drug: Chemotherapy; Radiation: Radiotherapy; Drug: blank placebo

INTERVENTIONS:
Procedure: Surgery — Maximum resection of the tumor (≥95%) with the help of conventional or intraoperative MRI neuronavigation. Confirmation will be proceeded by the contrast MRI within 72 hours after surgery.
Drug: Chemotherapy — Temozolomide(TMZ), 200mg·m^-2·d ×5 days，28 days every cycle. 6 cycles of TMZ are recommended.
Radiation: Radiotherapy — Standard dose, 4500 cGy to tumor with 3-cm margins, 1500 cGy boost to tumor bed.
Biological: DC vaccination — Eight to ten million dendritic cells (DCs) - administered via intradermal injections in 0.5 ml Phosphate Buffered Saline (PBS) in the shoulders near the back of the neck to facilitate trafficking of the DCs to the cervical lymph nodes.
  Arms: Arm DC
Drug: blank placebo — Saline that has the same appearance with DC vaccine.
  Arms: Arm Placebo

SUMMARY:
This is a Phase II study in a single center to determine the efficacy of autologous dendritic cells (DCs) loaded with autogeneic glioma stem-like cells (A2B5+) administered as a vaccination in adults with glioblastoma multiforme (primary or secondary).

DETAILED DESCRIPTION:
Despite the advances in diagnosis and treatment (surgery +radiation +chemotherapy), median survival for patients with newly diagnosed brain glioblastoma multiform (GBM) is about one year, for recurrent GBM is about 4 months. Recently, immunotherapy has emerged as a novel treatment strategy for glioma with improving patient survival. Usually, processed tumor antigens from the patient's own tumor or a peptide vaccine is capable of producing an anti-glioma response. Our previous experiment revealed that the CD133+ tumor stem-like cells associated antigens could elicit highly intensive immune response against human malignant glioma , and in phase I study, we have confirmed that DC vaccine loaded with glioma stem-like cells associated antigens against malignant glioma in recurrent patients was of safety .

Autologous DCs will be obtained from peripheral blood mononuclear cells (PBMCs) from each patient. Stem-like cells associated antigens (SAA) will be prepared with glioma stem-like cells that are harvested from patients with GBM and primary cultured and sorted flowcytometrically and then irradiated. Approximately 4 weeks will be required for vaccine production and the first vaccine administration. Each patient will receive an injection of DCs at his/her assigned dose once every week during the first 6 week. The dose of DCs is defined as 8~10×10^6.

Clinical trials that utilize DCs for immunotherapy have demonstrated significant survival benefit for patients who exhibit robust immune responses against tumor cells. Unfortunately, at the present time the majority of clinical trials were in phase I that illustrated the safety. The efficacy of DCs against glioblastoma is still lack of sufficient randomized phase II study. According to our previous phase I study, here we designed this clinical trial in a triple-blind randomized manner to validate the efficacy of DCs vaccination.

Recently，an exploratory randomized phase II clinical trial have been completed （Cancer immunology &immunotheapy ，2018，1677，1677-1688 ； PubMed ID: 30159779）， 43 GBM patients were randomized after surgery at a 1:1 ratio to receive either DCV (n = 22) or normal saline placebo (n = 21). Overall survival (OS) and progression-free survival (PFS) were analysed. Participants were stratified into different molecular subgroups based on the mutation (MT) status of isocitrate dehydrogenase (IDH1/2) and telomerase reverse transcriptase (TERT). Plasma cytokine levels, tumor-infiltrating lymphocyte numbers and immune co-inhibitory molecules PD-L1 and B7-H4 were also assessed. Multivariate Cox regression analysis revealed that DCV treatment significantly prolonged OS (p = 0.02) after adjusting for IDH1 and TERT promoter MT and B7-H4 expression, primary vs recurrent GBM. Among IDH1wild type (WT) TERTMT patients, DCV treatment significantly prolonged OS (p < 0.01) and PFS (p = 0.03) and increased plasma levels of cytokines CCL22 and IFN-γ compared with placebo. Patients with low B7-H4 expression showed significantly prolonged OS (p = 0.02) after DCV treatment.

In the present study, IDH1WTTERTMT subgroups of GBM patients more responsive to GSC DCV-based specific active-immunotherapy. However，It is noted that IDH1WTTERTMTGBM patients was analysed in a cohort samples which are not randomlized and the present study population is too small to evaluate conclusively demographic criteria for entry and patient recruitment. the results of the present study should be confirmed in a random cohort of IDH1WTTERTMT GBM patients. Accordingly , we made some modifications to the original plan, and are currently recruiting new participants.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed brain glioblastoma multiforme and molecular subgroups of IDH1 wildtype TERT mutation。
2. Patients with maximum safe resection of the tumor (≥95%) confirmed with contrast MR within 72 hours after surgery.
3. Age from 18 through 70 years.
4. Karnofsky performance score of ≥ 60%.
5. Adequate organ function within 14 days of study registration including the following:

   Adequate bone marrow reserve: absolute neutrophil (segmented and bands) count, (ANC) ≥ 1.0×10^9/L, platelets ≥100×10^9/L; hemoglobin ≥ 9 g/dL. Hepatic: bilirubin ≤1.3 mg/dL or 0-22 mmol/L, aspartate transaminase (AST) and alanine transaminase (ALT) < 3×upper limit of normal (ULN). Renal: Normal serum Creatinine for age (below) or creatinine clearance >60 ml/min/1.73 m^2. Electrocardiogram: normal.
6. Written informed consent must be obtained from all patients, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

1. Pregnant or breast-feeding patients. Pregnancy testing will be performed on all menstruating females within 14 days of study enrollment.
2. Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
3. Patients with history of immune system abnormalities such as hyperimmunity (e.g., autoimmune diseases) and hypoimmunity (e.g., myelodysplastic disorders, marrow failures, AIDS, ongoing pregnancy, transplant immuno-suppression), or medication of cortisol.
4. Patients with any conditions that could potentially alter immune function (e.g., AIDS, multiple sclerosis, diabetes, renal failure).
5. Patients currently received any other investigational agents.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-03 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) of the treatment using DC Vaccination for Glioblastoma with molecular markers for immunotherapy. | Every 4 weeks from baseline to 6 months.
  The objective response rate (ORR) is defined as the proportion of patients who achieve radiographic partial or complete response (PR or CR) according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 guideline.Molecular markers are based on the mutation (MT) status of isocitrate dehydrogenase (IDH1/2) and telomerase reverse transcriptase (TERT).

SECONDARY OUTCOMES:
Progression free survival | Every 4 weeks from baseline to 6 months.
  Progression free survival is defined as the time from the day in which the patient is enrolled to the date on which tumor progresses or the date on which the patient dies for any cause.
Overall survival | within 2 years after the surgery
  Overall survival is defined as the time from the day in which the patient is enrolled to the date on which the patient dies for any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Liangfu Zhou, M.D., Principal Investigator — Huashan Hospital
Locations (1):
- Huashan hospital, Fudan university, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Hua W, Yao Y, Chu Y, Zhong P, Sheng X, Xiao B, Wu J, Yang B, Mao Y, Zhou L. The CD133+ tumor stem-like cell-associated antigen may elicit highly intense immune responses against human malignant glioma. J Neurooncol. 2011 Nov;105(2):149-57. doi: 10.1007/s11060-011-0572-y. Epub 2011 Apr 11. PMID 21479962
- [Background] Hua Wei, Yao Yu, Chu Yiwei, Zhong Ping, Zhang Rong, Zhu Wei, Wu Jingsong, Ma Dexuan, Xu Ming, Mao Ying, Zhou Liangfu. Phase I study of dendritic cells pulsed with tumor stem-like cells associated antigens against malignant glioma in recurrent patients. Chinese Journal of Neurosurgery (Chinese). 2011, 27(1): 90-94.
- [Background] Xu M, Yao Y, Hua W, Wu Z, Zhong P, Mao Y, Zhou L, Luo F, Chu Y. Mouse glioma immunotherapy mediated by A2B5+ GL261 cell lysate-pulsed dendritic cells. J Neurooncol. 2014 Feb;116(3):497-504. doi: 10.1007/s11060-013-1334-9. Epub 2014 Jan 8. PMID 24398615
- [Background] Yao Y, Luo F, Tang C, Chen D, Qin Z, Hua W, Xu M, Zhong P, Yu S, Chen D, Ding X, Zhang Y, Zheng X, Yang J, Qian J, Deng Y, Hoon DSB, Hu J, Chu Y, Zhou L. Molecular subgroups and B7-H4 expression levels predict responses to dendritic cell vaccines in glioblastoma: an exploratory randomized phase II clinical trial. Cancer Immunol Immunother. 2018 Nov;67(11):1777-1788. doi: 10.1007/s00262-018-2232-y. Epub 2018 Aug 22. PMID 30159779